CLINICAL TRIAL: NCT00059215
Title: A Double-Blind, Randomized, Multicenter, Dose-Ranging Trial of CS-747 Compared With Clopidogrel in Subjects Undergoing Percutaneous Coronary Intervention
Brief Title: A Trial of CS-747 (Prasugrel) Compared With Clopidogrel in Patients Undergoing Percutaneous Coronary Intervention (PCI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7145; H7T-MC-TAAH (Other: Eli Lilly and Company)
Record Dates: First submitted 2003-04-21; First posted 2003-04-23 (Estimated); Results first posted 2010-05-21 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2010-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Prasugrel (CS-747) 40 mg LD/7.5 mg MD (Experimental): Prasugrel (CS-747) 40 mg oral loading dose (LD) at time of percutaneous coronary intervention (PCI) followed by 7.5 mg oral maintenance dose (MD), once daily, for 29-34 days
  Interventions: Drug: Prasugrel (CS-747)
- Prasugrel (CS-747) 60 mg LD/10 mg MD (Experimental): Prasugrel (CS-747) 60 mg oral loading dose (LD) at time of PCI followed by 10 mg oral maintenance dose (MD), once daily, for 29-34 days
  Interventions: Drug: Prasugrel (CS-747)
- Prasugrel (CS-747) 60 mg LD/15 mg MD (Experimental): Prasugrel (CS-747) 60 mg oral loading dose (LD) at time of PCI followed by 15 mg oral maintenance dose (MD), once daily, for 29-34 days
  Interventions: Drug: Prasugrel (CS-747)
- Clopidogrel (Active Comparator): Clopidogrel 300 mg oral LD at time of PCI followed by an oral 75 mg MD; taken once a day.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Prasugrel (CS-747) — Administered orally
  Other Names: Prasugrel; LY640315; Effient; Efient
  Arms: Prasugrel (CS-747) 40 mg LD/7.5 mg MD; Prasugrel (CS-747) 60 mg LD/10 mg MD; Prasugrel (CS-747) 60 mg LD/15 mg MD
Drug: Clopidogrel — Administered orally
  Arms: Clopidogrel

SUMMARY:
The purpose of this study is to evaluate the effects of a drug known as CS-747 (also known as prasugrel) on subjects having a procedure called a percutaneous coronary intervention (also referred to as PCI) in which a doctor will attempt to open a blocked vessel (or vessels) in the heart using a catheter (a long thin tube) that has a small balloon on the end. In many cases, patients who have this procedure receive a stent, a small wire spring that helps keep the vessel open.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be candidates for elective or urgent PCI with intended coronary stenting.
* Men or non-pregnant women (that is, postmenopausal women, women who are surgically sterile, or women of childbearing potential who have a negative urine or serum pregnancy test) who are greater than or equal to 18 and less than or equal to 75 years of age.

Exclusion Criteria:

* Patients must not have planned PCI procedure as initial treatment for an acute ST-elevation acute myocardial infarction (STEMI)
* Patients must not be receiving or will receive oral anticoagulation therapy that cannot be safely discontinued for the duration of the study
* Patients must not have cardiogenic shock or severe congestive heart failure
* Patients must not have active internal bleeding or history of bleeding diathesis
* Patients must not have prior history of hemorrhagic cerebrovascular accident (CVA) or nonhemorrhagic CVA within 2 years of enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 905 (Actual)
Dates: Start 2003-04; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Boston, Massachusetts, United States
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4599) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Victoria, British Columbia, Canada

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Prasugrel (CS-747) 40-mg LD/7.5 mg MD: Prasugrel (CS-747) 40 mg oral loading dose (LD) at time of percutaneous coronary intervention (PCI) followed by 7.5 mg oral maintenance dose (MD), once daily, for 29-34 days
- Prasugrel (CS-747) 60-mg LD/10-mg MD: Prasugrel (CS-747) 60-mg oral loading dose (LD) at time of PCI followed by 10-mg oral maintenance dose (MD), once daily, for 29-34 days
- Prasugrel (CS-747) 60-mg LD/15-mg MD: Prasugrel (CS-747) 60 mg oral loading dose (LD) at time of PCI followed by 15 mg oral maintenance dose (MD), once daily, for 29-34 days
Period: Overall Study
Arm/Group | Prasugrel (CS-747) 40-mg LD/7.5 mg MD | Prasugrel (CS-747) 60-mg LD/10-mg MD | Prasugrel (CS-747) 60-mg LD/15-mg MD | Clopidogrel
Started | 200 | 200 | 251 | 254
Completed | 187 (One subject discontinued before receiving treatment and is not included in the evaluable set.) | 186 | 236 | 239
Not Completed | 13 | 14 | 15 | 15
Not completed — Adverse Event | 5 | 5 | 9 | 9
Not completed — Death | 0 | 0 | 3 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 4 | 1 | 3
Not completed — Protocol Violation | 1 | 0 | 1 | 0
Not completed — Protocol entry criteria not met | 1 | 1 | 0 | 2
Not completed — Physician Decision | 1 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Prasugrel (CS-747) 40 mg LD/7.5 mg MD: Prasugrel (CS-747) 40-mg oral loading dose (LD) at time of percutaneous coronary intervention (PCI) followed by 7.5-mg oral maintenance dose (MD), once daily, for 29-34 days
- Prasugrel (CS-747) 60-mg LD/15-mg MD: Prasugrel (CS-747) 60-mg oral loading dose (LD) at time of PCI followed by 15-mg oral maintenance dose (MD), once daily, for 29-34 days
- Clopidogrel: Clopidogrel 300-mg oral LD at time of PCI followed by an oral 75-mg MD; taken once a day
- Total: Total of all reporting groups
Arm/Group | Prasugrel (CS-747) 40 mg LD/7.5 mg MD | Prasugrel (CS-747) 60 mg LD/10 mg MD | Prasugrel (CS-747) 60-mg LD/15-mg MD | Clopidogrel | Total
Number analyzed (Participants) | 199 | 200 | 251 | 254 | 904
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  >18 and <= 65 years | 129 | 152 | 185 | 195 | 661
  > 65 years | 70 | 48 | 66 | 59 | 243
Age Continuous [Mean (Standard Deviation); unit: years] | 60.4 (8.72) | 58.7 (9.15) | 59.4 (8.97) | 58.4 (9.17) | 59.2 (9.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 49 | 53 | 59 | 208
  Male | 152 | 151 | 198 | 195 | 696
Race/Ethnicity, Customized [Number; unit: participants]
  African descent | 10 | 14 | 15 | 9 | 48
  Western Asian | 3 | 3 | 1 | 3 | 10
  Caucasian | 180 | 180 | 226 | 238 | 824
  East/Southeast Asian | 1 | 1 | 1 | 0 | 3
  Hispanic | 5 | 2 | 7 | 2 | 16
  Other | 0 | 0 | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 43 | 44 | 48 | 46 | 181
  United States | 156 | 156 | 203 | 208 | 723

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-coronary Artery Bypass Graft (Non-CABG) Thrombolysis in Myocardial Infarction (TIMI) Major or Minor Bleeding Events
Description: Number of participants with non-coronary artery bypass graft (non-CABG) Thrombolysis In Myocardial Infarction (TIMI) Major or Minor bleeding.
  A major bleed was defined as an intracranial hemorrhage OR a clinically overt hemorrhage with a >5 g/dL decrease in hemoglobin.
  A minor bleed was defined as a clinically overt hemorrhage with a hemoglobin decrease >=3 g/dL and <= 5 g/dL.
Time Frame: randomization though 30 days after percutaneous coronary intervention (PCI)
Population: Patients who received at least one dose of study drug
Measure: Number; unit: participants
Groups:
- Prasugrel (CS-747) 40-mg LD/7.5-mg MD: Prasugrel (CS-747) 40-mg oral loading dose (LD) at time of PCI followed by 7.5 mg oral maintenance dose (MD), once daily, for 29-34 days
- Prasugrel (CS-747) 60-mg LD/10-mg MD: Prasugrel (CS-747) 60 mg oral loading dose (LD) at time of PCI followed by 10 mg oral maintenance dose (MD), once daily, for 29-34 days
- Prasugrel (CS-747) Combined: All evaluable patients in the 3 prasugrel (CS-747) treatment arms
Arm/Group | Prasugrel (CS-747) 40-mg LD/7.5-mg MD | Prasugrel (CS-747) 60-mg LD/10-mg MD | Prasugrel (CS-747) 60-mg LD/15-mg MD | Clopidogrel | Prasugrel (CS-747) Combined
Number analyzed (Participants) | 199 | 200 | 251 | 254 | 650
participants | 3 | 4 | 4 | 3 | 11
Statistical Analysis 1: Comparison: Prasugrel (CS-747) 40-mg LD/7.5-mg MD vs Prasugrel (CS-747) 60-mg LD/10-mg MD vs Prasugrel (CS-747) 60-mg LD/15-mg MD; Test type: Superiority or Other; p = 0.933, Fisher Exact
Statistical Analysis 2: Comparison: Clopidogrel vs Prasugrel (CS-747) Combined; Test type: Superiority or Other; p = 0.590, Log Rank

2. Secondary Outcome: Number of Participants With Major Adverse Cardiovascular Events (MACE)
Description: Number of participants with any of the following: death, nonfatal myocardial infarction, stroke, total or subtotal occlusion of the target vessel, urgent target vessel revascularization, recurrent ischemia requiring hospitalization.
Time Frame: randomization though 30 days after percutaneous coronary intervention (PCI)
Measure: Number; unit: participants
Arm/Group | Prasugrel (CS-747) 40-mg LD/7.5-mg MD | Prasugrel (CS-747) 60-mg LD/10-mg MD | Prasugrel (CS-747) 60-mg LD/15-mg MD | Clopidogrel | Prasugrel (CS-747) Combined
Number analyzed (Participants) | 199 | 200 | 251 | 254 | 650
participants | 15 | 15 | 17 | 24 | 47
Statistical Analysis 1: Comparison: Prasugrel (CS-747) 40-mg LD/7.5-mg MD vs Prasugrel (CS-747) 60-mg LD/10-mg MD vs Prasugrel (CS-747) 60-mg LD/15-mg MD; Test type: Superiority or Other; p = 0.945, Fisher Exact
Statistical Analysis 2: Comparison: Clopidogrel vs Prasugrel (CS-747) Combined; Test type: Superiority or Other; p = 0.260, Log Rank

3. Secondary Outcome: Number of Participants With Non-Coronary Artery Bypass Graft (Non-CABG) Thrombolysis in Myocardial Infarction (TIMI) Major Bleeding
Description: Number of participants with non-coronary artery bypass graft (non-CABG) Thrombolysis In Myocardial Infarction (TIMI) Major or Minor bleeding.
  A major bleed was defined as an intracranial hemorrhage OR a clinically overt hemorrhage with a >5 g/dL decrease in hemoglobin.
Time Frame: randomization though 30 days after percutaneous coronary intervention (PCI)
Measure: Number; unit: participants
Arm/Group | Prasugrel (CS-747) 40-mg LD/7.5-mg MD | Prasugrel (CS-747) 60-mg LD/10-mg MD | Prasugrel (CS-747) 60-mg LD/15-mg MD | Clopidogrel | Prasugrel (CS-747) Combined
Number analyzed (Participants) | 199 | 200 | 251 | 254 | 650
participants | 1 | 1 | 1 | 2 | 3
Statistical Analysis 1: Comparison: Prasugrel (CS-747) 40-mg LD/7.5-mg MD vs Prasugrel (CS-747) 60-mg LD/10-mg MD vs Prasugrel (CS-747) 60-mg LD/15-mg MD; Test type: Superiority or Other; p = 1.0, Fisher Exact
Statistical Analysis 2: Comparison: Clopidogrel vs Prasugrel (CS-747) Combined; Test type: Superiority or Other; p = 0.544, Log Rank

4. Secondary Outcome: Number of Participants With Non-CABG TIMI Major or Minor Bleeding Plus MACE
Description: Number of participants with non-coronary artery bypass graft (non-CABG) Thrombolysis In Myocardial Infarction (TIMI) Major or Minor bleeding or MACE.
  Major bleed was defined as an intracranial hemorrhage OR a clinically overt hemorrhage with a >5 g/dL decrease in hemoglobin.
  Minor bleed was defined as a clinically overt hemorrhage with a hemoglobin decrease >=3 g/dL and <= 5 g/dL.
  MACE is any of the following:death, nonfatal myocardial infarction, stroke, total or subtotal occlusion of the target vessel, urgent target vessel revascularization, recurrent ischemia requiring hospitalization
Time Frame: randomization though 30 days after percutaneous coronary intervention (PCI)
Measure: Number; unit: participants
Arm/Group | Prasugrel (CS-747) 40-mg LD/7.5-mg MD | Prasugrel (CS-747) 60-mg LD/10-mg MD | Prasugrel (CS-747) 60-mg LD/15-mg MD | Clopidogrel | Prasugrel (CS-747) Combined
Number analyzed (Participants) | 199 | 200 | 251 | 254 | 650
participants | 17 | 19 | 20 | 27 | 56
Statistical Analysis 1: Comparison: Clopidogrel vs Prasugrel (CS-747) Combined; Test type: Superiority or Other; p = 0.370, Fisher Exact

ADVERSE EVENTS:
Groups:
- Prasugrel (CS-747) 40-mg LD/7.5 mg MD: Prasugrel (CS-747) 40-mg oral loading dose (LD) at time of PCI followed by 7.5-mg oral maintenance dose (MD), once daily, for 29-34 days
- Prasugrel (CS-747) 60-mg LD/10 mg MD: Prasugrel (CS-747) 60-mg oral loading dose (LD) at time of PCI followed by 10-mg oral maintenance dose (MD), once daily, for 29-34 days
Arm/Group | Prasugrel (CS-747) 40-mg LD/7.5 mg MD | Prasugrel (CS-747) 60-mg LD/10 mg MD | Prasugrel (CS-747) 60-mg LD/15-mg MD | Clopidogrel
Serious Adverse Events (participants affected / at risk) | 17/199 | 9/200 | 18/251 | 22/254
Other Adverse Events (participants affected / at risk) | 147/199 | 157/200 | 192/251 | 195/254
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasugrel (CS-747) 40-mg LD/7.5 mg MD (N=199) | Prasugrel (CS-747) 60-mg LD/10 mg MD (N=200) | Prasugrel (CS-747) 60-mg LD/15-mg MD (N=251) | Clopidogrel (N=254)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia nos (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arterial haemorrhage nos (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood in stool (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac output decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site haemorrhage (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 6 (6) | 2 (2) | 6 (6) | 5 (5)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery dissection (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Coronary artery thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage nos (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia nos (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension nos (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemia nos (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Nodal rhythm (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scrotal haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasugrel (CS-747) 40-mg LD/7.5 mg MD (N=199) | Prasugrel (CS-747) 60-mg LD/10 mg MD (N=200) | Prasugrel (CS-747) 60-mg LD/15-mg MD (N=251) | Clopidogrel (N=254)
Angina pectoris (Cardiac disorders) | 18 (18) | 11 (11) | 15 (16) | 23 (25)
Anxiety (Psychiatric disorders) | 12 (12) | 7 (8) | 11 (11) | 15 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 19 (19) | 28 (28) | 28 (29)
Bradycardia nos (Cardiac disorders) | 5 (5) | 4 (4) | 16 (16) | 9 (10)
Catheter site discharge (General disorders) | 8 (9) | 13 (13) | 11 (11) | 8 (8)
Catheter site ecchymosis (General disorders) | 14 (14) | 15 (16) | 24 (24) | 12 (12)
Catheter site haemorrhage (General disorders) | 27 (29) | 35 (36) | 37 (39) | 30 (31)
Chest pain (General disorders) | 15 (15) | 21 (24) | 12 (12) | 19 (19)
Contusion (Skin and subcutaneous tissue disorders) | 9 (9) | 13 (16) | 20 (22) | 11 (12)
Dizziness (Nervous system disorders) | 11 (11) | 13 (13) | 12 (13) | 7 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 9 (11) | 14 (14) | 3 (3)
Headache (Nervous system disorders) | 9 (11) | 12 (12) | 17 (18) | 15 (15)
Hypertension nos (Vascular disorders) | 7 (7) | 11 (11) | 9 (9) | 8 (9)
Hypokalemia (Metabolism and nutrition disorders) | 10 (10) | 3 (3) | 9 (9) | 8 (8)
Hypotension nos (Vascular disorders) | 14 (14) | 11 (11) | 13 (13) | 17 (17)
Insomnia (Psychiatric disorders) | 8 (8) | 11 (11) | 11 (11) | 16 (16)
Nausea (Gastrointestinal disorders) | 18 (20) | 11 (11) | 23 (23) | 24 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days